CLINICAL TRIAL: NCT05428631
Title: Evaluation of the Tolerability and Safety of the CARDIOMEMS™ Intracardiac Continuous Cardiac Hemodynamic Monitoring Device in Patients with Cardio Renal Syndrome with Severe Renal Impairment
Brief Title: Tolerability and Safety of CARDIOMEMS™ Intracardiac Continuous Cardiac Hemodynamic Monitoring Device in Patients with Cardio Renal Syndrome with Severe Renal Impairment
Acronym: CARDIOMEMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: CHU Arnaud de Villeneuve MONTPELLIER (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AOI GCS-MERRI/2019/JER001
Record Dates: First submitted 2022-05-12; First posted 2022-06-23 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure; Renal Insufficiency
Keywords: Renal insufficiency,; heart failure,; medical device; blood pressure monitoring; tolerance
MeSH Terms: conditions — Heart Failure; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Patients will be pre-selected (pre-inclusion visit) during hospitalizations in the cardiology and nephrology departments of the Nîmes University Hospital. The study will be offered to any patient with class NYHA III heart failure who has been hospitalized in the previous 12 months for cardiac decompensation (current indication for the CARDIOMEMS™ system) and with advanced chronic renal failure with GFR (CKD-EPI) < 30 ml/min/1.73m2 persisting for more than 3 months and confirmed by Iohexol clearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CARDIOMEMS(TM) HF device (Experimental): Renal failure patients testing the CARDIOMEMS(TM) HF device
  Interventions: Device: Implantation of the CARDIOMEMS™ HF device

INTERVENTIONS:
Device: Implantation of the CARDIOMEMS™ HF device — The initial routine workup includes a nephrological evaluation: mGFR with Iohexol before fitting the CARDIOMEMS™ HF device, renal echo-Doppler, urinary sedimentation, etiological assessment of severe Chronic Kidney Disease, NT-ProBNP, impedancemetry, urinary ionogram, weight, anemia assessment, and correction of possible iron and/or vitamin deficiency and a cardiology evaluation: blood pressure, heart rate, clinical data, biology (Complete Blood Count, iono, urea, creatinine, total bilirubin, ferritin, CST), echocardiography (Left Ventricle Ejection Fraction, E/A, E/e', indexed volume of the left atrium, Tricuspid Annular Plane Systolic Excursion, Tissue Doppler S-wave, surface area of the right atrium, Systolic Pulmonary Artery Pressure, Right Atrial Pressure). The device will be implanted in the selected patients by Pr François Roubille at Montpellier University Hospital within 1 month of the pre-inclusion visit. It will monitor their pulmonary artery pressure.
  Other Names: Nephrolocical evaluation measured with the CARDIOMEMS™ HF device

SUMMARY:
Renal failure is present in 40% of heart failure patients, and is one of the main comorbidities of heart failure. Follow-up with pulmonary artery pressure (PAP) monitoring has shown a reduction in mortality and frequency of hospitalization in patients with heart failure alone in the CHAMPION trial. Patients with New York Heart Association class III heart failure and a hospitalization in the previous 12 months were included in that study. They benefited from the "CardioMEMS™ HF" device with a sensor implanted in the pulmonary artery to measure PAP. According to that study, the information led to more precise and early adaptation of therapy by avoiding the onset of heart failure symptoms and reducing the number of hospitalizations. However, in that study, patients with impaired renal function (Glomerular Filtration Rate<25 mL/min/1.73m2) were excluded, limiting the indication for treatment in those patients, and the evolution of renal function during the study was not reported.

Patients with heart failure AND advanced renal failure are defined as having a cardio-renal syndrome, with strong interaction between these 2 organs. In the event of predominant right heart failure, they may require treatment by renal replacement or dialysis. There seems to be a link between high venous pressure, renal repercussions and the need for dialysis. Additional follow-up data in this clinical situation are needed to confirm this link and to suggest the interest of continuous PAP monitoring to improve the management of these patients with cardio-renal syndrome with severe renal impairment defined by a Glomerular Filtration Rate< 30 ml/min/1.73m2 (KDIGO Cardio-renal 2019). This pilot study aims to evaluate how tolerable the "CARDIOMEMS™ HF" device in patients with cardio-renal syndrome and obtain the first information on the relationship between cardiac hemodynamics and renal function in this population.

DETAILED DESCRIPTION:
There are currently 1.5 million heart failure patients in France. The high morbidity and mortality make it a major public health issue. Renal failure, present in 40% of these patients, is one of the main comorbidities of heart failure and makes its management more complex. Medical follow-up with pulmonary artery pressure (PAP) monitoring has shown a reduction in mortality and frequency of hospitalization in patients with heart failure alone in the CHAMPION trial. Patients with New York Heart Association class III heart failure and a hospitalization in the previous 12 months were included in this study. They benefited from the "CardioMEMS™ HF" device with implantation of a sensor in the pulmonary artery allowing direct and continuous measurement of PAP. According to this study, this information allowed for more precise and early adaptation of therapy by avoiding the occurrence of heart failure symptoms and reducing the frequency of hospitalizations. In this study, patients with impaired renal function were excluded (Glomerular Filtration Rate <25 mL/min/1.73m2), limiting the indication for treatment in these patients, and the evolution of renal function during the study was not reported.

Patients with heart failure associated with advanced renal failure are defined as having a cardio-renal syndrome, with a strong interaction between these 2 organs that may, in particular in the case of predominant right heart failure, require treatment by renal replacement or dialysis. According to the data available to date, the predominant hypothesis is a link between high venous pressure, renal repercussions and the need for dialysis. Additional follow-up data in this clinical situation are needed to confirm this link and to suggest the interest of continuous monitoring of PAP to improve the management of these patients with cardio-renal syndrome with severe renal impairment defined by a Glomerular Filtration Rate< 30 ml/min/1.73m2 (KDIGO Cardio-renal 2019). Therefore, the investigators wish to initiate a pilot study evaluating the tolerability of the "CARDIOMEMS™ HF" device in patients with cardio renal syndrome and obtain the first information on the relationship between cardiac hemodynamics and renal function in this population.

This is the first pilot study on the safety and tolerability of the use of the CardioMEMS™ HF medical device in cardio renal syndrome with severe renal impairment (documented by Glomerular Filtration Rate < 30 mL/min/1.73m2 measured by Iohexol clearance) treated medically and without renal replacement therapy.

In this study, the CARDIOMEMS™ HF device, the most successful implanted pulmonary arterial pressure monitoring system currently available on the market will be implemented. Its teletransmitted information can guide the treatment of patients with heart failure.This system, by responding to the recent international recommendations which advocate a better understanding of the hemodynamic situation in this pathology with in particular the link between pulmonary arterial pressure and renal function, could help us to identify innovative evaluation tools with a view to improving therapeutic management with the new treatments available in heart failure (AA House et al: HF in kidney disease: a KDIGO conference report).

ELIGIBILITY:
Inclusion Criteria:

* Patient with class NYHA III heart failure having been hospitalized in the previous 12 months for cardiac decompensation (the current indication for the CARDIOMEMS™ system), right heart failure or biventricular heart failure with the definition of TAPSE<15mm and/or SDTI<9.5cm/s regardless of LVEF, NtproBNP>1500 pg/ml.
* Patient with advanced renal failure with GFR (CKD-EPI) < 30 ml/min/1.73m2 for more than 3 months confirmed by GFR measurement (Iohexol clearance)
* Patient with a pulmonary artery greater than 7 mm in diameter.
* The patient has been informed of the study set-up, objectives, constraints and patient rights.
* The patient must have given free and informed consent and signed the consent form.
* The patient must be affiliated or a beneficiary of a health insurance plan. Precautions: if the patient is on anticoagulant therapy, an International Normalized Ratio <1.5 is recommended before right heart catheterization and any implantation procedure

Exclusion Criteria:

* Patients with a contraindication to the CARDIOMEMS™ HF system (pulmonary embolism with sequelae, artery less than 7 mm, active infection).
* Patients already on renal replacement therapy.
* Patients with a history of acute venous thrombosis.
* Patients unable to tolerate right heart catheterization.
* Patients with a major cardiovascular event (i.e., myocardial infarction, stroke) within 2 months of the initial examination.
* Patients with congenital heart disease or mechanical right heart valve(s).
* Patients with known hypersensitivity or allergy to aspirin and/or clopidogrel.
* Patients with a body mass index >35. Measure the patient's chest circumference at the armpit: if the patient's chest circumference is > 165 cm, the sensor should not be implanted.
* Patients unable to take dual anti-platelet therapy or anticoagulant therapy for one month after implantation
* Patient hypersensitive or allergic to iohexol.
* Patient is participating in another Class I interventional study, or has participated in another interventional study within the last 3 months.
* Patient is in an exclusion period determined by a previous study.
* Patient is under guardianship, conservatorship, or conservatorship.
* The patient refuses to sign the consent form.
* It is impossible to give the patient informed information.
* The patient is pregnant or nursing.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2026-08-26 (Estimated); Study Completion 2027-08-26 (Estimated)

PRIMARY OUTCOMES:
Adverse events | On the day of implanting the Cardiomems device
  Perioperative collection of complications related to the puncture site (hematoma, arteriovenous fistula) and right catheterization (arrhythmia, peri-procedure heart failure decompensation).
Adverse events | One month after implanting the Cardiomems device
  Monthly collection of adverse events over the 12-month follow-up period. In particular, cardiac parameters will be collected (sensor failure, migration, re-calibration, re-intervention, gas embolism, allergic reaction, abnormal heart rate or rhythm, bleeding, hematoma, chest pain, nausea, vascular accident, infection, sepsis, delayed healing, atrial dysrhythmia clot formation, ecchymosis, vascular trauma, valve damage, pulmonary infarction, pulmonary embolism, heart attack (myocardial infarction), death, hemoptysis, separation of sensor and delivery system impossible) and renal (risk of infection, thrombotic risk, interference with dialysis catheter placement).
Adverse events | Two months after implanting the Cardiomems device
  Perioperative collection of complications related to the puncture site (hematoma, arteriovenous fistula) and right catheterization (arrhythmia, peri-procedure heart failure decompensation).
  Monthly collection of adverse events over the 12-month follow-up period. In particular, cardiac parameters will be collected (sensor failure, migration, re-calibration, re-intervention, gas embolism, allergic reaction, abnormal heart rate or rhythm, bleeding, hematoma, chest pain, nausea, vascular accident, infection, sepsis, delayed healing, atrial dysrhythmia clot formation, ecchymosis, vascular trauma, valve damage, pulmonary infarction, pulmonary embolism, heart attack (myocardial infarction), death, hemoptysis, separation of sensor and delivery system impossible) and renal (risk of infection, thrombotic risk, interference with dialysis catheter placement).
Adverse events | Three months after implanting the Cardiomems device
  Monthly collection of adverse events over the 12-month follow-up period. In particular, cardiac parameters will be collected (sensor failure, migration, re-calibration, re-intervention, gas embolism, allergic reaction, abnormal heart rate or rhythm, bleeding, hematoma, chest pain, nausea, vascular accident, infection, sepsis, delayed healing, atrial dysrhythmia clot formation, ecchymosis, vascular trauma, valve damage, pulmonary infarction, pulmonary embolism, heart attack (myocardial infarction), death, hemoptysis, separation of sensor and delivery system impossible) and renal (risk of infection, thrombotic risk, interference with dialysis catheter placement).
Adverse events | Four months after implanting the Cardiomems device
  Monthly collection of adverse events over the 12-month follow-up period. In particular, cardiac parameters will be collected (sensor failure, migration, re-calibration, re-intervention, gas embolism, allergic reaction, abnormal heart rate or rhythm, bleeding, hematoma, chest pain, nausea, vascular accident, infection, sepsis, delayed healing, atrial dysrhythmia clot formation, ecchymosis, vascular trauma, valve damage, pulmonary infarction, pulmonary embolism, heart attack (myocardial infarction), death, hemoptysis, separation of sensor and delivery system impossible) and renal (risk of infection, thrombotic risk, interference with dialysis catheter placement).
Adverse events | Five months after implanting the Cardiomems device
  Monthly collection of adverse events over the 12-month follow-up period. In particular, cardiac parameters will be collected (sensor failure, migration, re-calibration, re-intervention, gas embolism, allergic reaction, abnormal heart rate or rhythm, bleeding, hematoma, chest pain, nausea, vascular accident, infection, sepsis, delayed healing, atrial dysrhythmia clot formation, ecchymosis, vascular trauma, valve damage, pulmonary infarction, pulmonary embolism, heart attack (myocardial infarction), death, hemoptysis, separation of sensor and delivery system impossible) and renal (risk of infection, thrombotic risk, interference with dialysis catheter placement).
Adverse events | Six months after implanting the Cardiomems device
  Monthly collection of adverse events over the 12-month follow-up period. In particular, cardiac parameters will be collected (sensor failure, migration, re-calibration, re-intervention, gas embolism, allergic reaction, abnormal heart rate or rhythm, bleeding, hematoma, chest pain, nausea, vascular accident, infection, sepsis, delayed healing, atrial dysrhythmia clot formation, ecchymosis, vascular trauma, valve damage, pulmonary infarction, pulmonary embolism, heart attack (myocardial infarction), death, hemoptysis, separation of sensor and delivery system impossible) and renal (risk of infection, thrombotic risk, interference with dialysis catheter placement).
Adverse events | Seven months after implanting the Cardiomems device
  Monthly collection of adverse events over the 12-month follow-up period. In particular, cardiac parameters will be collected (sensor failure, migration, re-calibration, re-intervention, gas embolism, allergic reaction, abnormal heart rate or rhythm, bleeding, hematoma, chest pain, nausea, vascular accident, infection, sepsis, delayed healing, atrial dysrhythmia clot formation, ecchymosis, vascular trauma, valve damage, pulmonary infarction, pulmonary embolism, heart attack (myocardial infarction), death, hemoptysis, separation of sensor and delivery system impossible) and renal (risk of infection, thrombotic risk, interference with dialysis catheter placement).
Adverse events | Eight months after implanting the Cardiomems device
  Monthly collection of adverse events over the 12-month follow-up period. In particular, cardiac parameters will be collected (sensor failure, migration, re-calibration, re-intervention, gas embolism, allergic reaction, abnormal heart rate or rhythm, bleeding, hematoma, chest pain, nausea, vascular accident, infection, sepsis, delayed healing, atrial dysrhythmia clot formation, ecchymosis, vascular trauma, valve damage, pulmonary infarction, pulmonary embolism, heart attack (myocardial infarction), death, hemoptysis, separation of sensor and delivery system impossible) and renal (risk of infection, thrombotic risk, interference with dialysis catheter placement).
Adverse events | Nine months after implanting the Cardiomems device
  Monthly collection of adverse events over the 12-month follow-up period. In particular, cardiac parameters will be collected (sensor failure, migration, re-calibration, re-intervention, gas embolism, allergic reaction, abnormal heart rate or rhythm, bleeding, hematoma, chest pain, nausea, vascular accident, infection, sepsis, delayed healing, atrial dysrhythmia clot formation, ecchymosis, vascular trauma, valve damage, pulmonary infarction, pulmonary embolism, heart attack (myocardial infarction), death, hemoptysis, separation of sensor and delivery system impossible) and renal (risk of infection, thrombotic risk, interference with dialysis catheter placement).
Adverse events | Ten months after implanting the Cardiomems device
  Monthly collection of adverse events over the 12-month follow-up period. In particular, cardiac parameters will be collected (sensor failure, migration, re-calibration, re-intervention, gas embolism, allergic reaction, abnormal heart rate or rhythm, bleeding, hematoma, chest pain, nausea, vascular accident, infection, sepsis, delayed healing, atrial dysrhythmia clot formation, ecchymosis, vascular trauma, valve damage, pulmonary infarction, pulmonary embolism, heart attack (myocardial infarction), death, hemoptysis, separation of sensor and delivery system impossible) and renal (risk of infection, thrombotic risk, interference with dialysis catheter placement).
Adverse events | Eleven months after implanting the Cardiomems device
  Monthly collection of adverse events over the 12-month follow-up period. In particular, cardiac parameters will be collected (sensor failure, migration, re-calibration, re-intervention, gas embolism, allergic reaction, abnormal heart rate or rhythm, bleeding, hematoma, chest pain, nausea, vascular accident, infection, sepsis, delayed healing, atrial dysrhythmia clot formation, ecchymosis, vascular trauma, valve damage, pulmonary infarction, pulmonary embolism, heart attack (myocardial infarction), death, hemoptysis, separation of sensor and delivery system impossible) and renal (risk of infection, thrombotic risk, interference with dialysis catheter placement).
Adverse events | Twelve months after implanting the Cardiomems device
  Monthly collection of adverse events over the 12-month follow-up period. In particular, cardiac parameters will be collected (sensor failure, migration, re-calibration, re-intervention, gas embolism, allergic reaction, abnormal heart rate or rhythm, bleeding, hematoma, chest pain, nausea, vascular accident, infection, sepsis, delayed healing, atrial dysrhythmia clot formation, ecchymosis, vascular trauma, valve damage, pulmonary infarction, pulmonary embolism, heart attack (myocardial infarction), death, hemoptysis, separation of sensor and delivery system impossible) and renal (risk of infection, thrombotic risk, interference with dialysis catheter placement).

SECONDARY OUTCOMES:
Estimated effect on renal function | Between 1 day to 1 month before implanting the device.
  The estimated Glomerular Filtration Rate (eGFR) will be recorded in mL/min
Measured effect on renal function | Between 1 day to 1 month before implanting the device.
  The Glomerular Filtration Rate measured with Iohexol (mGFR) will be recorded in mL/min.
Estimated effect on renal function | Day 0 (day of implanting the device)
  The estimated Glomerular Filtration Rate (eGFR) will be recorded in mL/min
Measured effect on renal function | Day 0 (day of implanting the device)
  The Glomerular Filtration Rate measured with Iohexol (mGFR) will be recorded in mL/min.
Estimated effect on renal function | Month 3
  The estimated Glomerular Filtration Rate (eGFR) will be recorded in mL/min
Measured effect on renal function | Month 3
  The Glomerular Filtration Rate measured with Iohexol (mGFR) will be recorded in mL/min.
Estimated effect on renal function | Month 6
  The estimated Glomerular Filtration Rate (eGFR) will be recorded in mL/min
Measured effect on renal function | Month 6
  The Glomerular Filtration Rate measured with Iohexol (mGFR) will be recorded in mL/min.
Estimated effect on renal function | Month 9
  The estimated Glomerular Filtration Rate (eGFR) will be recorded in mL/min
Measured effect on renal function | Month 9
  The Glomerular Filtration Rate measured with Iohexol (mGFR) will be recorded in mL/min.
Estimated effect on renal function | Month 12
  The estimated Glomerular Filtration Rate (eGFR) will be recorded in mL/min.
Measured effect on renal function | Month 12
  The Glomerular Filtration Rate measured with Iohexol (mGFR) will be recorded in mL/min.
Re-hospitalizations | Month 12
  Any re-hospitalizations will be recorded for a period of up to 12 months of follow-up
Vital status | Month 12
  Patient dead or alive
Link between cardiac hemodynamics and renal function: Pulmonary Arterial Pressure | From Day 0 (day of implanting the device) to the end of Month 12
  Pulmonary Arterial Pressure will be continuously monitored for 12 months by the CardioMEMS™ HF intracardiac device in patients with severe cardio-renal syndrome and measured in Hg.
Link between cardiac hemodynamics and renal function: Glomerular Filtration Rate | Day 0
  Glomerular Filtration Rate will be measured by measuring plasma clearance of iohexol from a single sample.
Link between cardiac hemodynamics and renal function: Pulmonary Arterial Pressure | Month 3
  Pulmonary Arterial Pressure will be continuously monitored for 12 months by the CardioMEMS™ HF intracardiac device in patients with severe cardio-renal syndrome and measured in Hg. Readings will be recorded at 3-monthly intervals.
Link between cardiac hemodynamics and renal function: Glomerular Filtration Rate | Month 3
  Glomerular Filtration Rate will be measured in ml/min/1.72² by measuring plasma clearance of iohexol from a single sample.
Link between cardiac hemodynamics and renal function: Pulmonary Arterial Pressure | Month 6
  Pulmonary Arterial Pressure will be continuously monitored for 12 months by the CardioMEMS™ HF intracardiac device in patients with severe cardio-renal syndrome and measured in Hg. Readings will be recorded at 3-monthly intervals.
Link between cardiac hemodynamics and renal function: Glomerular Filtration Rate | Month 6
  Glomerular Filtration Rate will be measured in ml/min/1.72² by measuring plasma clearance of iohexol from a single sample.
Link between cardiac hemodynamics and renal function: Pulmonary Arterial Pressure | Month 9
  Pulmonary Arterial Pressure will be continuously monitored for 12 months by the CardioMEMS™ HF intracardiac device in patients with severe cardio-renal syndrome and measured in Hg. Readings will be recorded at 3-monthly intervals.
Link between cardiac hemodynamics and renal function: Glomerular Filtration Rate | Month 9
  Glomerular Filtration Rate will be measured in ml/min/1.72² by measuring plasma clearance of iohexol from a single sample.
Link between cardiac hemodynamics and renal function: Pulmonary Arterial Pressure | Month 12
  Pulmonary Arterial Pressure will be continuously monitored for 12 months by the CardioMEMS™ HF intracardiac device in patients with severe cardio-renal syndrome and measured in Hg. Readings will be recorded at 3-monthly intervals.
Link between cardiac hemodynamics and renal function: Glomerular Filtration Rate | Month 12
  Glomerular Filtration Rate will be measured in ml/min/1.72² by measuring plasma clearance of iohexol from a single sample.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: exertional dyspnea | Day 0
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  To quantify dyspnea, the patient is asked to indicate on a visual analog scale the point corresponding to his/her own perception, evaluated as the distance from the zero extreme (non dyspnea) and expressed as a percentage of the total length of the line.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: exertional dyspnea | Month 3
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  To quantify dyspnea, the patient is asked to indicate on a visual analog scale the point corresponding to his/her own perception, evaluated as the distance from the zero extreme (non dyspnea) and expressed as a percentage of the total length of the line.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: exertional dyspnea | Month 6
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  To quantify dyspnea, the patient is asked to indicate on a visual analog scale the point corresponding to his/her own perception, evaluated as the distance from the zero extreme (non dyspnea) and expressed as a percentage of the total length of the line.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: exertional dyspnea | Month 9
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  To quantify dyspnea, the patient is asked to indicate on a visual analog scale the point corresponding to his/her own perception, evaluated as the distance from the zero extreme (non dyspnea) and expressed as a percentage of the total length of the line.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: exertional dyspnea | Month 12
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  To quantify dyspnea, the patient is asked to indicate on a visual analog scale the point corresponding to his/her own perception, evaluated as the distance from the zero extreme (non dyspnea) and expressed as a percentage of the total length of the line.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: NT-pro-BNP biomarkers | Day 0
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form. Natriuretic Peptide Tests (BNP, NT-proBNP) will be made on a single blood sample. BNP and NT-proBNP will be measured as percentages.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: NT-pro-BNP biomarkers | Month 3
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form. Natriuretic Peptide Tests (BNP, NT-proBNP) will be made on a single blood sample. BNP and NT-proBNP will be measured in %.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: NT-pro-BNP biomarkers | Month 6
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form. Natriuretic Peptide Tests (BNP, NT-proBNP) will be made on a single blood sample. BNP and NT-proBNP will be measured as percentages.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: NT-pro-BNP biomarkers | Month 9
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form. Natriuretic Peptide Tests (BNP, NT-proBNP) will be made on a single blood sample. BNP and NT-proBNP will be measured as percentages.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: NT-pro-BNP biomarkers | Month 12
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form. Natriuretic Peptide Tests (BNP, NT-proBNP) will be made on a single blood sample. BNP and NT-proBNP will be measured as percentages.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: left ventricular ejection fraction | Day 0
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Left Ventricular Ejection Fraction will be measured as a percentage via the formula EF=SV/EDV (ejection fraction = stroke volume/end diastolic volume.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: left ventricular ejection fraction | Month 3
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Left Ventricular Ejection Fraction will be measured as a percentage via the formula EF=SV/EDV (ejection fraction = stroke volume/end diastolic volume.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: left ventricular ejection fraction | Month 6
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Left Ventricular Ejection Fraction will be measured as a percentage via the formula EF=SV/EDV (ejection fraction = stroke volume/end diastolic volume.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: left ventricular ejection fraction | Month 9
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Left Ventricular Ejection Fraction will be measured as a percentage via the formula EF=SV/EDV (ejection fraction = stroke volume/end diastolic volume.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: left ventricular ejection fraction | Month 12
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Left Ventricular Ejection Fraction will be measured as a percentage via the formula EF=SV/EDV (ejection fraction = stroke volume/end diastolic volume.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: E/A | Month 0
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  E/A will be measured as a ratio.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: E/A | Month 3
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  E/A will be measured as a ratio (the E/A ratio is the ratio of the early (E) to late (A) ventricular filling velocities).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: E/A | Month 6
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  E/A will be measured as a ratio (the E/A ratio is the ratio of the early (E) to late (A) ventricular filling velocities).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: E/A | Month 9
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  E/A will be measured as a ratio (the E/A ratio is the ratio of the early (E) to late (A) ventricular filling velocities).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: E/A | Month 12
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  E/A will be measured as a ratio (the E/A ratio is the ratio of the early (E) to late (A) ventricular filling velocities).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: E/e' | Month 0
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form. E/e' will be measured as a ratio.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: E/e' | Month 3
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form. E/e' will be measured as a ratio (E= early diastolic transmitral flow velocity and e' = early diastolic mitral annular velocity).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: E/e' | Month 6
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form. E/e' will be measured as a ratio (E= early diastolic transmitral flow velocity and e' = early diastolic mitral annular velocity).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: E/e' | Month 9
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form. E/e' will be measured as a ratio (E= early diastolic transmitral flow velocity and e' = early diastolic mitral annular velocity).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: E/e' | Month 12
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form. E/e' will be measured as a ratio (E= early diastolic transmitral flow velocity and e' = early diastolic mitral annular velocity).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Indexed left atrial volume | Month 0
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Indexed left atrial volume will be measured in ml/m2.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Indexed left atrial volume | Month 3
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Indexed left atrial volume will be measured in ml/m2.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Indexed left atrial volume | Month 6
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Indexed left atrial volume will be measured in ml/m2.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Indexed left atrial volume | Month 9
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Indexed left atrial volume will be measured in ml/m2.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Indexed left atrial volume | Month 12
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Indexed left atrial volume will be measured in ml/m2.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Tricuspid Annular Plane Systolic Excursion | Month 0
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Tricuspid Annular Plane Systolic Excursion will be measured in cm.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Tricuspid Annular Plane Systolic Excursion | Month 3
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Tricuspid Annular Plane Systolic Excursion will be measured in cm.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Tricuspid Annular Plane Systolic Excursion | Month 6
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Tricuspid Annular Plane Systolic Excursion will be measured in cm.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Tricuspid Annular Plane Systolic Excursion | Month 9
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Tricuspid Annular Plane Systolic Excursion will be measured in cm.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Tricuspid Annular Plane Systolic Excursion | Month 12
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Tricuspid Annular Plane Systolic Excursion will be measured in cm.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Tissue Doppler S-wave | Month 0
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Tissue Doppler S-wave will be measured in mV
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Tissue Doppler S-wave | Month 3
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Tissue Doppler S-wave will be measured in mV
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Tissue Doppler S-wave | Month 6
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Tissue Doppler S-wave will be measured in mV
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Tissue Doppler S-wave | Month 9
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Tissue Doppler S-wave will be measured in mV
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Tissue Doppler S-wave | Month 12
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Tissue Doppler S-wave will be measured in mV
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Right atrium area | Month 0
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Right atrium area will be measured in cm2.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Right atrium area | Month 3
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Right atrium area will be measured in cm2.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Right atrium area | Month 6
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Right atrium area will be measured in cm2.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Right atrium area | Month 9
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Right atrium area will be measured in cm2.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Right atrium area | Month 12
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Right atrium area will be measured in cm2.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Systolic pulmonary artery pressure | Month 0
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Systolic pulmonary artery pressure will be measured in mmHg.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Systolic pulmonary artery pressure | Month 3
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Systolic pulmonary artery pressure will be measured in mmHg.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Systolic pulmonary artery pressure | Month 6
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Systolic pulmonary artery pressure will be measured in mmHg.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Systolic pulmonary artery pressure | Month 9
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Systolic pulmonary artery pressure will be measured in mmHg.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Systolic pulmonary artery pressure | Month 12
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Systolic pulmonary artery pressure will be measured in mmHg.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Right atrial pressure | Month 0
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Right atrial pressure will be measured in mmHg.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Right atrial pressure | Month 3
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Right atrial pressure will be measured in mmHg.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Right atrial pressure | Month 6
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Right atrial pressure will be measured in mmHg.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Right atrial pressure | Month 9
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Right atrial pressure will be measured in mmHg.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Right atrial pressure | Month 12
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Right atrial pressure will be measured in mmHg.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Stroke volume | Day 0
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Stroke volume (SV) will be measured and recorded in millilitres per square metre (ml/m2).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Stroke volume | Month 3
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Stroke volume (SV) will be measured and recorded in millilitres per square metre (ml/m2).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Stroke volume | Month 6
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Stroke volume (SV) will be measured and recorded in millilitres per square metre (ml/m2).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Stroke volume | Month 9
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Stroke volume (SV) will be measured and recorded in millilitres per square metre (ml/m2).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Stroke volume | Month 12
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form. Stroke volume (SV) will be measured and recorded in millilitres per square metre (ml/m2).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Heart rate | Day 0
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form. The patient's heart rate (HR) will be measured and recorded as beats per minute (BPM).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Heart rate | Month 3
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form. The patient's heart rate (HR) will be measured and recorded as beats per minute (BPM).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Heart rate | Month 6
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form. The patient's heart rate (HR) will be measured and recorded as beats per minute (BPM).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Heart rate | Month 9
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form. The patient's heart rate (HR) will be measured and recorded as beats per minute (BPM).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: Heart rate | Month 12
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form. The patient's heart rate (HR) will be measured and recorded as beats per minute (BPM).
Comparison of cardiac hemodynamic monitoring data with the clinical picture: cardiac output | Day 0
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Cardiac output (CO) will be measured and recorded in liters per minute.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: cardiac output | Month 3
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Cardiac output (CO) will be measured and recorded in liters per minute.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: cardiac output | Month 6
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Cardiac output (CO) will be measured and recorded in liters per minute.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: cardiac output | Month 9
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Cardiac output (CO) will be measured and recorded in liters per minute.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: cardiac output | Month 12
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Cardiac output (CO) will be measured and recorded in liters per minute.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: ventricular ejection time | Day 0
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Ventricular ejection time (VET) will be measured and recorded in milliseconds.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: ventricular ejection time | Month 3
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Ventricular ejection time (VET) will be measured and recorded in milliseconds.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: ventricular ejection time | Month 6
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Ventricular ejection time (VET) will be measured and recorded in milliseconds.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: ventricular ejection time | Month 9
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Ventricular ejection time (VET) will be measured and recorded in milliseconds.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: ventricular ejection time | Month 12
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Ventricular ejection time (VET) will be measured and recorded in milliseconds.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: pre-ejection period | Day 0
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Stroke volume (SV), heart rate (HR), cardiac output (CO) ventricular ejection time (VET) and pre-ejection period (PER) will all be measured and recorded in milliseconds.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: pre-ejection period | Month 3
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Stroke volume (SV), heart rate (HR), cardiac output (CO) ventricular ejection time (VET) and pre-ejection period (PER) will all be measured and recorded in milliseconds.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: pre-ejection period | Month 6
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Stroke volume (SV), heart rate (HR), cardiac output (CO) ventricular ejection time (VET) and pre-ejection period (PER) will all be measured and recorded in milliseconds.
Comparison of cardiac hemodynamic monitoring data with the clinical picture: pre-ejection period | Month 9
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Stroke volume (SV), heart rate (HR), cardiac output (CO) ventricular ejection time (VET) and pre-ejection period (PER) will all be measured and recorded in milliseconds .
Comparison of cardiac hemodynamic monitoring data with the clinical picture: pre-ejection period | Month 12
  The cardiac hemodynamic monitoring data will be compared with the clinical picture (exertional dyspnea, peak VO2 max) and currently available assessment tools (NT-pro-BNP biomarkers, echocardiography, impedancemetry) recorded in the electronic case report form.
  Stroke volume (SV), heart rate (HR), cardiac output (CO) ventricular ejection time (VET) and pre-ejection period (PER) will all be measured and recorded in milliseconds.
Patient quality of life | Day 0
  The patient's quality of life will be evaluated using the EQ-5D questionnaire. This questionnaire essentially consists of two pages: the EQ-5D descriptive system (page 2 of the questionnaire) and the EQ-5D visual analog scale (EQ VAS) (page 3 of the questionnaire) ranging from 0 - 100 in which 0 = extremely bad health and 100 = excellent health.
  EQ-5D is not an abbreviation and is the correct term to use when referring to the instrument.
  The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression.
Patient quality of life | Month 3
  The patient's quality of life will be evaluated using the EQ-5D questionnaire. This questionnaire essentially consists of two pages: the EQ-5D descriptive system (page 2 of the questionnaire) and the EQ-5D visual analog scale (EQ VAS) (page 3 of the questionnaire) ranging from 0 - 100 in which 0 = extremely bad health and 100 = excellent health.
  EQ-5D is not an abbreviation and is the correct term to use when referring to the instrument.
  The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression.
Patient quality of life | Month 6
  The patient's quality of life will be evaluated using the EQ-5D questionnaire. This questionnaire essentially consists of two pages: the EQ-5D descriptive system (page 2 of the questionnaire) and the EQ-5D visual analog scale (EQ VAS) (page 3 of the questionnaire) ranging from 0 - 100 in which 0 = extremely bad health and 100 = excellent health.
  EQ-5D is not an abbreviation and is the correct term to use when referring to the instrument.
  The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression.
Patient quality of life | Month 9
  The patient's quality of life will be evaluated using the EQ-5D questionnaire. This questionnaire essentially consists of two pages: the EQ-5D descriptive system (page 2 of the questionnaire) and the EQ-5D visual analog scale (EQ VAS) (page 3 of the questionnaire) ranging from 0 - 100 in which 0 = extremely bad health and 100 = excellent health.
  EQ-5D is not an abbreviation and is the correct term to use when referring to the instrument.
  The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression.
Patient quality of life | Month 12
  The patient's quality of life will be evaluated using the EQ-5D questionnaire. This questionnaire essentially consists of two pages: the EQ-5D descriptive system (page 2 of the questionnaire) and the EQ-5D visual analog scale (EQ VAS) (page 3 of the questionnaire).
  EQ-5D is not an abbreviation and is the correct term to use when referring to the instrument.
  The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression.
  The EQ -5D is scored from 0 -100 and the VAS is scored from 0 -10.

OTHER OUTCOMES:
Age of patients | Day 0
  In years
Weight of patients | Day 0
  In kilograms
Height of patients | Day 0
  In centimeters
Patient's cardiac history | Day 0
  The type of cardiopathy (ischemic, rhythmic, valvular, primitive dilated, hypertrophic, toxic, restrictive etc; will all be recorded.
Cardiovascular risk factors | Day 0
  All cardiovascular risk factors such as smoking, high blood pressure, diabetes, dyslipidemia, overweight, chronic inflammatory disease, family background, sleep apnea syndrome , etc. will all be recorded.
Cardiac devices | Day 0
  Any devices such as a Pacemaker, defibrillator, resynchronization etc. will all be recorded.
Etiology of renal disease | Day 0
  The etiology of renal disease will be described and recorded.
Renal history | Day 0
  The patient's previous renal function (information from the patient's medical file) will be recorded.
Medication received | Day 0
  All medication received, especially medication for heart failure: ACEI/sartan, beta-blockers, ARM, sacubitril-valsartan will be recorded.
Diuretics received | Day 0
  All loop diuretics in equivalent dose of furosemide and thiazide diuretics and antialdosterone will be recorded together with their dosages.
Iron supplementation received | Day 0
  Any iron supplementation received will be recorded together with the dosage.
Transferrin | Month 6
  mg/dL
Transferrin | Month 12
  mg/dL
Ferritin | Month 6
  ng/ mL
Ferritin | Month 12
  ng/ mL

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Etienne RICCI, Dr., Principal Investigator — Nîmes University Hospital; François ROUBILLE, Prof., Principal Investigator — CHU Arnaud de Villeneuve MONTPELLIER; Guillaume CAYLA, Prof., Principal Investigator — Nîmes University Hospital; Sylvain AGUILHON, Dr., Principal Investigator — CHU Arnaud de Villeneuve MONTPELLIER; Sylvain CARIOU, Dr., Principal Investigator — Nîmes University Hospital
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard
  - CHRU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier

IPD SHARING:
Plan to Share IPD: No